CLINICAL TRIAL: NCT05555589
Title: A Phase 3, Multi-Center, Randomized, Parallel, Double Masked, Placebo-Controlled Clinical Study to Assess the Safety and Efficacy of 0.1% RGN-259 Ophthalmic Solution for the Treatment of Neurotrophic Keratopathy (SEER-2)
Brief Title: Assessment of the Safety and Efficacy of 0.1% RGN-259 Ophthalmic Solution for the Treatment of NK: SEER-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ReGenTree, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-NK-302
Record Dates: First submitted 2022-09-15; First posted 2022-09-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Neurotrophic Keratopathy
Keywords: Neurotrophic Keratitis; NK
MeSH Terms: interventions — thymosin beta(4)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.1% RGN-259 Opthalmic Solution (Experimental): It is a preservative-free, sterile eye drop solution containing Tβ4 for direct instillation into study eye(s), five times per day for 28 days
  Interventions: Drug: RGN-259
- Placebo Ophthalmic Solution (Vehicle for RGN-259 Ophthalmic Solution) (Placebo Comparator): It is composed of the same excipients as RGN-259 but does not contain Tβ4
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RGN-259 — A preservative-free, sterile eye drop solution containing Tβ4 for direct instillation into study eye(s), five times per day for 28 days
  Other Names: Tβ4; Thymosin Beta 4; Timbetasin
  Arms: 0.1% RGN-259 Opthalmic Solution
Drug: Placebo — It is composed of the same excipients as RGN-259 but does not contain Tβ4. Direct instillation into study eye(s), five times per day for 28 days
  Other Names: Vehicle Control
  Arms: Placebo Ophthalmic Solution (Vehicle for RGN-259 Ophthalmic Solution)

SUMMARY:
The objective of this study is to compare the safety and efficacy of RGN-259 to placebo for the treatment of Neurotrophic Keratopathy (NK)

DETAILED DESCRIPTION:
Neurotrophic keratopathy (NK) is a degenerative corneal disease that occurs as a result of partial or total impairment of trigeminal innervation. The resulting loss of corneal sensitivity (anesthesia) leads to a reduction in lacrimation and a decline in status, metabolism, and mitosis of corneal epithelial cells.

ELIGIBILITY:
Inclusion Criteria

1. Be male or female of any race, at least 18 years of age;
2. Have provided written informed consent;
3. Be able and willing to follow instructions, including participation in all study assessments and visits;
4. At the time of Visit 1, have documentation or observation of a Persistent Epithelial Defect (PED) in one or both eyes, defined as a corneal epithelial defect that has not resolved after 1 week of conventional treatment using non-preserved ocular lubricants, non-preserved topical ophthalmic antibiotics, oral doxycycline, patching, amniotic membrane, serum tears, and/or therapeutic contact lenses;
5. Have stage 2 or 3 neurotrophic keratopathy (Mackie Classification) in at least one eye of which the longest dimension (length or width) of the defect measures a minimum length of 1 mm (study eye) and which is confirmed by the Investigator not to be simply superficial punctate keratitis, at Visit 1;
6. Have evidence of decreased corneal sensitivity ≤40 mm using the Cochet-Bonnet aesthesiometer at Visit 1;
7. Have BCVA score ≤75 letter counts in the study eye based on the ETDRS protocol;
8. Have at least one eye (the same eye) satisfy all criteria for d, e, f, g above;
9. Female subjects of child-bearing potential must be non-lactating and using and agree to continue using an acceptable method of contraception for at least 4 weeks prior to the first dose of study product and until 12 weeks after last dose, and have a negative urine pregnancy test during screening;
10. Male subjects must agree to use an adequate method of contraception.

Exclusion Criteria

1. Have any condition that, in the opinion of the Investigator, would interfere with the subject's ability to complete the study, would interfere with the interpretation of safety or efficacy, or would present an undue risk to the subject.
2. Have any clinically significant slit-lamp findings in the study eye that in the opinion of the Investigator may interfere with the study parameters;
3. Clinically significant active blepharitis, meibomian gland dysfunction (MGD), or lid margin inflammation, or active ocular allergy in study eye that requires treatment that in the opinion of the investigator may interfere with the study parameters;
4. Have a Unanesthetized Schirmer's test score of ≤3 mm at Visit 1;
5. Have a lid function abnormality (ex. Lagophthalmos) which, in the opinion of the Investigator, is the primary cause of the persistent epithelial defect;
6. Have an ongoing ocular infection (bacterial, viral or fungal) or active inflammation (e.g., follicular conjunctivitis) in the study eye.
7. History of any ocular surgery (including laser or refractive surgical procedures) within the three months before study enrollment.
8. Prior surgical procedure(s) for the treatment of NK (e.g., tarsorrhaphy, conjunctival flap, etc.) within the three months before study enrollment with the exception of amniotic membrane transplantation.
9. Have any planned ocular surgical procedures or are likely to require ocular surgery for the study eye during the study;
10. Have received Botox® injection to induce blepharoptosis in the study eye within 90 days prior to Visit 1;
11. Have used contact lenses (for therapeutic or refractive correction) in the study eye within 14 days prior to Visit 1, or anticipate use of contact lenses during the study period.
12. Have used OxervateTM in the study eye within the past 2 months;
13. Anticipate use of serum tears in the study eye during the study period.
14. Have a presence or history of any ocular or systemic disorder or condition that might hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the Investigator to be incompatible with the study visit schedule or conduct;
15. Have used drugs which affect lacrimation or function of the trigeminal nerve within 30 days of Visit 1 or anticipate use of these systemic medication throughout the course of the study;
16. Have any autoimmune or chronic inflammatory disease that might have hindered the efficacy of the study treatment or its evaluation;
17. Be on topical (Ocular/Nasal) immunosuppressive therapy within 30 days prior to screening or is likely to require this during the course of the study;
18. Have a known allergy and/or sensitivity to the study product or its components;
19. History of drug, medication or alcohol abuse or addiction;
20. Have participated in an investigational drug study within 30 days prior to screening;
21. Have fever, inflammation, or systemic signs of illness suggestive of systemic or invasive infection, including COVID-19 or a positive test for COVID-19, within 2 weeks prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects achieving complete healing of PED at Day 29 | Day 29
  Percentage of subjects achieving complete healing of the Persistent Epithelial Defect (PED) at Day 29 determined by corneal fluorescein staining as measured by the Central Reading Center.

SECONDARY OUTCOMES:
Percentage of subjects achieving complete healing of PED at Day 29 | Day 29
  Percentage of subjects achieving complete healing of the PED determined by corneal fluorescein staining as measured by the Investigator.
Percentage change from baseline of lesion size | Day 8, 15, 22, 29, 36, and 43
  Percentage change from baseline of lesion size determined by corneal fluorescein staining (measurements of greatest dimension of fluorescein staining)
NK stage by Mackie classification | Day 8, 15, 22, 29, 36, and 43
  NK stage graded according to the Mackie classification (Stage I, II, III. Higher scores mean a better or worse outcome)
Visual Acuity determined by ETDRS | Day 8, 15, 22, 29, 36, and 43
  Visual Acuity determined by Early Treatment of Diabetic Retinopathy Study (ETDRS)
Corneal sensitivity inside the lesion determined by Cochet Bonnet aesthesiometer (Unit: mm) | Day 8, 15, 22, 29, 36, and 43

OTHER OUTCOMES:
Frequency and severity of AEs | Day 8, 15, 22, 29, 36, and 43
  Frequency and severity of AEs as reported according to the NCI CTCAE version 5.0
Number of participants with abnormal vital signs | Day 1, 8, 15, 22, 29, 36, and 43
  Blood pressure, heart rate, respiratory rate, oxygen saturation, and body temperature will be measured and assessed its clinical abnormality.
Intraocular Pressure (Unit: mmHg) | Day 1, 8, 29 and 43
Dilated fundoscopy (Vitreous, Retina, Macula, Choroid, Optic Nerve) | Day 1, 8, 29 and 43
  The fundoscopy exam will be performed and clinical abnormality of vitreous, retina, Macula, Choroid and Optic Nerve will be described.
Slit-lamp biomicroscopy (Cornea, Conjunctiva, Anterior Chamber, Iris, Lens, Lid) | Day 1, 8, 15, 22, 29, 36, and 43
  The Slit-Lamp biomicroscopy will be performed and clinical abnormality of Cornea, Conjunctiva, Anterior Chamber, Iris, Lens and Lid will be described.

CONTACTS AND LOCATIONS:
Locations (36):
- United States (29):
  - Harvard Eye Associates, Laguna Hills, California
  - Loma Linda University Eye Institute, Loma Linda, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Advance Vision Research Institute, Longmont, Colorado
  - Connecticut Eye Consultants, P.C. Danbury Eye Physicians & Surgeons, Danbury, Connecticut
  - Nature Coast Clinical Research, Crystal River, Florida
  - University of Miami - Bascom Palmer Eye Institute, Miami, Miami, Florida
  - University of South Florida, Ophthalmolgoy, Tampa, Florida
  - Thomas Eye Group, P.C., Sandy Springs, Georgia
  - Northwestern, Chicago, Illinois
  - Midwest Cornea Associates, LLC., Carmel, Indiana
  - Huffman & Huffman, PSC, Lexington, Kentucky
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Washington University Eye Center, St Louis, Missouri
  - Metropolitan Eye Research and Surgery Institute, Palisades Park, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Duke Eye Center, Durham, North Carolina
  - Oculus Research, Raleigh, North Carolina
  - CORE, Inc. / Vita Eye Clinic, Shelby, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cole Eye Institute, Cleveland, Ohio
  - Pacific ClearVision Institute, Eugene, Oregon
  - Cataract & Laser Institute of Southern Oregon, Medford, Oregon
  - OHSU Casey Eye Institute, Portland, Oregon
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - MCOA Eye Care, San Antonio, Texas
  - Berkeley Eye Center, Sugar Land, Texas
  - Virginia Eye Consultants, Norfolk, Virginia
  - University of Washington, Department of Ophthalmology, Seatle, Washington
- Italy (2):
  - Università di Brescia, Brescia, Brescia
  - Azienda Ospedaliero Universitaria Careggi, Florence, Firenze
- Gabinet Okulistyczny Prof Edward Wylegala, Katowice, Silesian Voivodeship, Poland
- Spain (4):
  - IMO Barcelona, Grupo Miranza, Barcelona, Barcelona
  - Hospital La Arruzafa, Córdoba, Córdoba
  - Instituto Oftalmológico Fernández-Vega, Oviedo, Principality of Asturias
  - Aiken Prevención & Cirugía Ocular, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No